CLINICAL TRIAL: NCT00033488
Title: The UK Familial Ovarian Cancer Screening Study
Brief Title: Screening Women at High Genetic Risk for Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000069292; UKFOCSS; CRCA-FOCS; EU-20044
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-06

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Other: cytology specimen collection procedure
Procedure: annual screening
Procedure: comparison of screening methods

SUMMARY:
RATIONALE: Screening tests may help doctors detect cancer cells early and plan more effective treatment for ovarian cancer.

PURPOSE: Screening trial to determine the best procedure to detect ovarian cancer in women who have a high genetic risk for developing ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine an optimal screening procedure for ovarian cancer, in terms of the most appropriate screening test, criteria for interpretation of results, and screening intervals, in women at high genetic risk for developing ovarian cancer.
* Determine the physical morbidity and the resource implications associated with ovarian cancer screening in these women.
* Assess the feasibility of screening this high-risk population in terms of compliance rates.

OUTLINE: Patients undergo transvaginal ultrasonography of the ovaries (scheduled for the early follicular phase, day 3-6 of the menstrual cycle) and CA 125 measurement annually. Blood samples are collected every 4 months for analysis of CA 125 levels and novel markers.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 5,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* First-degree relative (mother, sister, or daughter) of an affected member of a high-risk family defined as one of the following:

  * Family containing 2 or more individuals with ovarian cancer who are connected by first-degree relationships
  * Family containing 1 individual with ovarian cancer and 1 individual with breast cancer and under 50 years of age at the time of diagnosis who are connected by first-degree relationships
  * Family containing 1 individual with ovarian cancer and 2 individuals with breast cancer and under 60 years of age at the time of diagnosis who are connected by first-degree relationships
  * Family containing an affected individual with a mutation of one of the known ovarian cancer predisposing genes
  * Family containing 3 individuals with colorectal cancer with at least 1 individual under 50 years of age at time of diagnosis and 1 individual with ovarian cancer who are connected by first-degree relationships
  * Families where affected relatives are related by second-degree relationships through an unaffected intervening male relative who has an affected daughter are allowed

PATIENT CHARACTERISTICS:

Age:

* 35 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* No prior bilateral oophorectomy

Other:

* No concurrent participation in other ovarian cancer screening trials

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2000-09; Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Mackay, MD, MA, FRCP, FRCPE, Study Chair — Institute of Child Health
Locations (2):
- United Kingdom (2):
  - Saint Bartholomew's Hospital, London, England
  - Institute of Child Health, London, England